CLINICAL TRIAL: NCT05549986
Title: Discriminant Ability of the Shock Index, Modified Shock Index, and Reverse Shock Index Multiplied by the Glasgow Coma Scale on Mortality in Adult Trauma Patients: A PATOS Study
Status: Completed | Type: Observational
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Tse-Hao Chen, Principal Investigator, Mackay Memorial Hospital
Other Study IDs: 21MMHIS389e
Record Dates: First submitted 2022-08-29; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Trauma; Shock, Traumatic; Morality
Keywords: Shock index(SI); Modified Shock Index (MSI); Reverse Shock Index Multiplied by the Glasgow Coma Scale (rSIG); Mortality; Pan-Asian Trauma Outcomes Study (PATOS)
MeSH Terms: conditions — Wounds and Injuries; Shock, Traumatic | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mortality group: Patients encountered in-hospital mortality or 30-day mortality
  Interventions: Other: Observational
- Survival group: Patients did not encounter in-hospital mortality or 30-day mortality
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational

SUMMARY:
We evaluated a cohort of adult trauma patients transported to emergency departments. The first vital signs were used to calculate the SI, MSI, and rSIG. The areas under the receiver operating characteristic curves (AUROCs) and test results were used to compare the discriminant performance of the indices on short-term mortality and poor functional outcome. A subgroup analysis of geriatric patients, traumatic brain injury, penetrating injury, and non-penetrating injury was performed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) EMS-transported from January 2016 to December 2020

Exclusion Criteria:

* Patients with missing entries of age, sex, triage, SBP, DBP, HR, or GCS were excluded.
* Entries with missing records of in-hospital mortality or 30-day mortality were excluded from the short-term mortality cohort analyses.
* Patients without a Modified Rankin Scale (MRS) record at discharge were excluded from the functional outcome cohort analyses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study included adult patients (≥18 years) EMS-transported from January 2016 to December 2020. Patients with missing entries of age, sex, triage, SBP, DBP, HR, or GCS were excluded. Entries with missing records of in-hospital mortality or 30-day mortality were excluded from the short-term mortality cohort analyses. Patients without a Modified Rankin Scale (MRS) record at discharge were excluded from the functional outcome cohort analyses.
Sampling Method: Non-Probability Sample
Enrollment: 105641 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Discriminant power of SI, MSI, and rSIG on short-term mortality for adult traumatic patients | 30 days
  AUROC in associated with short-term mortality with SI, MSI, rSIG

SECONDARY OUTCOMES:
Discriminant power of SI, MSI, and rSIG on functional outcome for adult traumatic patients | We defined no symptoms, no significant disability, slight disability, and moderate disability (MRS 0-3) as favorable functional outcomes and moderately severe disability, severe disability, and death (MRS 4-6) as poor functional outcomes
  AUROC in associated with functional outcome with SI, MSI, rSIG

CONTACTS AND LOCATIONS:
Overall Officials: Tse-Hao Chen, M.D., Principal Investigator — Mackay Memorial Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen TH, Wu MY, Do Shin S, Jamaluddin SF, Son DN, Hong KJ, Jen-Tang S, Tanaka H, Hsiao CH, Hsieh SL, Chien DK, Tsai W, Chang WH, Chiang WC; PATOS Clinical Research Network. Discriminant ability of the shock index, modified shock index, and reverse shock index multiplied by the Glasgow coma scale on mortality in adult trauma patients: a PATOS retrospective cohort study. Int J Surg. 2023 May 1;109(5):1231-1238. doi: 10.1097/JS9.0000000000000287. PMID 37222717